CLINICAL TRIAL: NCT01169363
Title: Validation of AML Proteomic Signature Associated With Clinical Response to Ara-C Based Induction Therapy in Patients 60 Years of Age or Older Using Samples From ECOG Studies 3999, 3993 and 1490
Brief Title: Biomarkers in Bone Marrow and Blood Samples From Older Patients With Acute Myeloid Leukemia Treated With Cytarabine-Based Therapy
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000681533; ECOG-E1L09T1
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: proteomic profiling
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of bone marrow and blood from patients with cancer in the laboratory may help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is studying biomarkers in bone marrow and blood samples from older patients with acute myeloid leukemia treated with cytarabine-based therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To validate a pre-specified proteomic classifier to predict the likelihood of complete response (CR) to cytarabine-based induction chemotherapy in older patients with non-M3 acute myeloid leukemia.

Secondary

* To identify signaling nodes associated with risk of relapse among these patients who achieve a CR to induction chemotherapy.

OUTLINE: This is a multicenter study.

Previously collected bone marrow and peripheral blood samples are analyzed to validate the association of a pre-specified proteomic signature with clinical response via flow cytometry.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Treated on EST-1490, E-3993, or ECOG-E3999
* Bone marrow and peripheral blood samples collected at diagnosis and before induction chemotherapy available
* No M3 disease

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients enrolled on E3999 and E3993 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-07-08 (Actual); Primary Completion 2010-08-08 (Actual); Study Completion 2010-08-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving a complete response to induction chemotherapy | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Paietta, PhD, Principal Investigator — Our Lady of Mercy Medical Center